CLINICAL TRIAL: NCT04536194
Title: Hemodynamic Effects of Dopamine Versus Norepinephrine Under General Anesthesia in Infant With Congenital Heart Disease
Brief Title: Dopamine Versus Norepinephrine Under General Anesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Zhijian Zhou, vice director of department of anesthesiology, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mzk-0003-2020
Record Dates: First submitted 2020-08-21; First posted 2020-09-02 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Anesthesia; Infant; Congenital Heart Disease; Hemodynamic Instability
Keywords: norepinephrine; dopamine
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Norepinephrine; Dopamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- norepinephrine (Experimental): infusion of norepinephrine with a adjusted dose to elevate 10% of mean arterial pressure
  Interventions: Drug: norepinephrine
- Dopamine (Active Comparator): infusion of dopamine with a adjusted dose to elevate 10% of mean arterial pressure
  Interventions: Drug: dopamine

INTERVENTIONS:
Drug: norepinephrine — to treat hypotension under general anesthesia with norepinephrine
  Arms: norepinephrine
Drug: dopamine — to treat hypotension under general anesthesia with dopamine
  Arms: Dopamine

SUMMARY:
Participants under general anesthesia will be randomly treated with an adjusted dose dopamine or norepinephrine to elevate 10% of mean arterial pressure. Systemic hemodynamic data is recorded by PRAM and the change of cardiac index is compared between groups.

DETAILED DESCRIPTION:
After intubation under general anesthesia, radial arterial is cannulated and pressure transducer is connected to MostCare(core technique PRAM). CI, SVRI, SVI, SVV, dp/dt and HR are recorded before and after a infusion of dopamine or norepinephrine to elevate 10% of mean arterial pressure. Changes of these hemodynamic data are compared.

ELIGIBILITY:
Inclusion Criteria:

* undertake cardiac surgery for congenital heart disease

Exclusion Criteria:

* Aortic valve or aortic disease
* severe arrhythmia
* use of cardiovascular active drugs before anesthesia
* need to use a combination of different cardiovascular support drugs after anesthesia

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
changes of cardiac index | 20 minutes
  the differences of cardiac index between after and before the intervention (l/min/m2)

SECONDARY OUTCOMES:
changes of stroke volume index | 20 minutes
  the differences of stroke volume index between after and before the intervention (ml/m2)
changes of systemic vascular resistance index | 20 minutes
  the differences of systemic vascular resistance index between after and before the intervention(dyne ∙ sec ∙ m2/cm5)
changes of the maximal slope of systolic upstroke | 20 minutes
  the differences of the maximal slope of systolic upstroke between after and before the intervention(mmHg/ms)
changes of heart rate | 20 minutes
  the differences of heart rate between after and before the intervention (bpm)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 6 months after publication
Access Criteria: share to researchers by email

REFERENCES:
- [Background] Yuan SM. Acute kidney injury after pediatric cardiac surgery. Pediatr Neonatol. 2019 Feb;60(1):3-11. doi: 10.1016/j.pedneo.2018.03.007. Epub 2018 Mar 30. PMID 29891225
- [Background] Foulon P, De Backer D. The hemodynamic effects of norepinephrine: far more than an increase in blood pressure! Ann Transl Med. 2018 Nov;6(Suppl 1):S25. doi: 10.21037/atm.2018.09.27. No abstract available. PMID 30613600
- [Background] Cavigelli-Brunner A, Hug MI, Dave H, Baenziger O, Buerki C, Bettex D, Cannizzaro V, Balmer C. Prevention of Low Cardiac Output Syndrome After Pediatric Cardiac Surgery: A Double-Blind Randomized Clinical Pilot Study Comparing Dobutamine and Milrinone. Pediatr Crit Care Med. 2018 Jul;19(7):619-625. doi: 10.1097/PCC.0000000000001533. PMID 29538053
- [Background] Saxena R, Durward A, Steeley S, Murdoch IA, Tibby SM. Predicting fluid responsiveness in 100 critically ill children: the effect of baseline contractility. Intensive Care Med. 2015 Dec;41(12):2161-9. doi: 10.1007/s00134-015-4075-8. Epub 2015 Sep 28. PMID 26415680
- [Result] Hamzaoui O, Jozwiak M, Geffriaud T, Sztrymf B, Prat D, Jacobs F, Monnet X, Trouiller P, Richard C, Teboul JL. Norepinephrine exerts an inotropic effect during the early phase of human septic shock. Br J Anaesth. 2018 Mar;120(3):517-524. doi: 10.1016/j.bja.2017.11.065. Epub 2017 Nov 21. PMID 29452808
- [Result] Favia I, Rizza A, Garisto C, Haiberger R, Di Chiara L, Romagnoli S, Ricci Z. Cardiac index assessment by the pressure recording analytical method in infants after paediatric cardiac surgery: a pilot retrospective study. Interact Cardiovasc Thorac Surg. 2016 Dec;23(6):919-923. doi: 10.1093/icvts/ivw251. Epub 2016 Aug 1. PMID 27481679
- [Result] Urbano J, Lopez J, Gonzalez R, Solana MJ, Fernandez SN, Bellon JM, Lopez-Herce J. Measurement of cardiac output in children by pressure-recording analytical method. Pediatr Cardiol. 2015 Feb;36(2):358-64. doi: 10.1007/s00246-014-1014-3. Epub 2014 Sep 2. PMID 25179459
- [Result] Garisto C, Favia I, Ricci Z, Romagnoli S, Haiberger R, Polito A, Cogo P. Pressure recording analytical method and bioreactance for stroke volume index monitoring during pediatric cardiac surgery. Paediatr Anaesth. 2015 Feb;25(2):143-9. doi: 10.1111/pan.12360. Epub 2014 Feb 3. PMID 24491036